CLINICAL TRIAL: NCT05588609
Title: A Phase 2 Study Evaluating Activity of Zenocutuzumab (MCLA-128) in Patients With or Without Molecularly Defined Cancers
Brief Title: Study Evaluating Zenocutuzumab in Patients With or Without Molecularly Defined Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Merus terminated the study early due to changes in organizational priorities.
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-128-CL03
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: NSCLC Harboring NRG1 Fusion; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Afatinib; enzalutamide; Abiraterone Acetate; zenocutuzumab

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: NSCLC harboring NRG1+ fusion (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab once every 2 weeks in combination with afatinib 40 mg orally once daily.
  Interventions: Drug: Afatinib Oral Tablet; Biological: MCLA-128
- Part 1: mCRPC (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab once every 2 weeks in combination with the AR targeting agent they experienced disease progression on prior to study entry:
  enzalutamide 160 mg orally once daily or abiraterone 1000 mg orally once daily with prednisone 5 mg orally twice daily.
  Interventions: Drug: Enzalutamide Pill; Drug: Abiraterone acetate tablets; Biological: MCLA-128
- Part 2: NSCLC harboring NRG1+ fusion (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab once every 2 weeks in combination with afatinib 40 mg orally once daily.
  Interventions: Drug: Afatinib Oral Tablet; Biological: MCLA-128
- Part 2: mCRPC (Experimental): Participants will receive intravenous infusion of 750 mg of zenocutuzumab once every 2 weeks in combination with the AR targeting agent they experienced disease progression on prior to study entry:
  enzalutamide 160 mg orally once daily or abiraterone 1000 mg orally once daily with prednisone 5 mg orally twice daily
  Interventions: Drug: Enzalutamide Pill; Drug: Abiraterone acetate tablets; Biological: MCLA-128

INTERVENTIONS:
Drug: Afatinib Oral Tablet — anti epidermal growth factor receptor (EGFR)/HER2 agent
  Other Names: GILOTRIF®; GIOTRIF®
  Arms: Part 1: NSCLC harboring NRG1+ fusion; Part 2: NSCLC harboring NRG1+ fusion
Drug: Enzalutamide Pill — second-generation androgen receptor antagonist
  Other Names: XTANDI®
  Arms: Part 1: mCRPC; Part 2: mCRPC
Drug: Abiraterone acetate tablets — androgen synthesis inhibitor
  Other Names: ZYTIGA®
  Arms: Part 1: mCRPC; Part 2: mCRPC
Biological: MCLA-128 — full length IgG1 bispecific antibody targeting HER2 and HER3
  Other Names: Zenocutuzumab

SUMMARY:
This is a Phase II, open-label, 2-arm, multicenter, international study designed to evaluate the efficacy of zenocutuzumab alone or in combination in patients with the following diagnoses:

Group A: NRG1+ NSCLC Group B: mCRPC

DETAILED DESCRIPTION:
Study Design:

This is an open label (all participants know the identity of the study drug), multicenter (more than one study site), study consisting of 2 parts:

Group A (NRG1+ NSCLC): Approximately 50 NRG1+NSCLC patients will be enrolled and will receive zenocutuzumab in combination with afatinib 40 mg orally once daily.

Group B (mCRPC): Up to 40 mCRPC patients will be enrolled and will receive zenocutuzumab in combination with the AR targeting agent enzalutamide or abiraterone on which they experienced disease progression immediately before study entry.

For the administration of zenocutuzumab in combination in Groups A and B, the Treatment Period will include 2 phases, an initial safety run-in phase, and an expansion phase with an interim efficacy analysis.

The study will consist of 4 periods: Screening, Treatment, Safety Follow-up, and Long-term Follow up.

ELIGIBILITY:
Inclusion Criteria: (Groups A, B)

1. Signed informed consent before initiation of any study procedures.
2. Age ≥ 18 years at signature of informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Estimated life expectancy of ≥ 12 weeks.
5. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA).
6. Adequate organ function:

   * Absolute neutrophil count ≥ 1.5 × 109/L.
   * Hemoglobin ≥ 9 g/dL.
   * Platelets ≥ 100 × 109/L.
   * Serum calcium within normal ranges (or corrected with supplements).
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (in case of liver involvement by malignancy, ALT/AST ≤ 5 × ULN will be allowed).
   * Total bilirubin ≤ 1.5 × ULN (in case of Gilbert disease, total bilirubin ≤ 3 × ULN will be allowed).
   * Estimated glomerular filtration rate of > 30 mL/min based on the Cockroft-Gault formula (Appendix D).
   * Serum albumin > 3.0 g/dL.
7. Availability of a representative tumor specimen, either a formalin-fixed paraffin embedded (FFPE) de novo (ie, obtained up to 2 months before signing of the informed consent form [ICF]) or an FFPE archival tumor sample, preferably collected within 2 years of the start of study treatment. A fresh FFPE sample is preferred.
8. Sexually active male and female patients of childbearing potential must agree to use contraceptive measures.

Inclusion Criteria: (Group A Only)

A1. Have histologically confirmed locally advanced, unresectable, or metastatic NSCLC harboring an NRG1 gene fusion detected by DNA- or RNA-based next generation sequencing in a tumor sample or in plasma-cell free DNA. A2. Have received prior standard therapy appropriate for the tumor type and disease or must be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy in the opinion of the Investigator or have no satisfactory available treatment options. A3. Have at least 1 measurable lesion per RECIST v1.1. A4. Able to swallow oral medications and absence of gastrointestinal conditions (eg, malabsorption, resection) deemed to jeopardize intestinal absorption.

Inclusion Criteria: (Group B Only) B1. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features. B2. Metastatic disease documented by at least 2 bone lesions on whole body bone scintigraphy, or soft tissue disease documented by computed tomography (CT) scan/magnetic resonance imaging (MRI). B3. Ongoing androgen deprivation with a serum testosterone level ≤ 1.73 nmol/L (≤ 50 ng/dL) at Screening. B4. Current ongoing therapy with a next-generation AR signaling inhibitor (enzalutamide or abiraterone) started at least 90 days before Screening. B5. Progressive disease by PCWG3 criteria B6. Able to swallow oral medications and absence of gastrointestinal conditions (eg, malabsorption, resection) deemed to jeopardize intestinal absorption.

Exclusion Criteria: (Groups A, B)

1. Central nervous system metastases that are untreated or symptomatic, or require radiation, surgery, or continued steroid therapy to control symptoms within 14 days of study entry.
2. Previous exposure to anti-HER3-directed therapies.
3. Known leptomeningeal involvement.
4. Participation in another interventional clinical trial or treatment with any investigational drug within 4 weeks before study entry.
5. Chronic use of high-dose oral corticosteroid therapy (> 10 mg of prednisone- equivalent a day).
6. Uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) or unstable angina.
7. History of congestive heart failure Class II-IV by New York Heart Association criteria, or serious cardiac arrhythmia requiring treatment (except atrial fibrillation, or paroxysmal supraventricular tachycardia).
8. History of myocardial infarction within 6 months of study entry.
9. History of prior or concomitant malignancies (other than excised nonmelanoma skin cancer, cured in situ cervical carcinoma, or low-grade Ta or T1 urothelial carcinoma of the bladder that has undergone potentially curative therapy) within 3 years of study entry.
10. Current serious illness or medical conditions including, but not limited to uncontrolled active infection, and clinically significant pulmonary, metabolic, or psychiatric disorders.
11. Patients with the following known infectious diseases:

    * Known active hepatitis B infection (hepatitis B surface antigen [HBsAg] positive) without receiving antiviral treatment.
    * Known positive test for hepatitis C virus (HCV) RNA.
12. Known human immunodeficiency virus (HIV)-positive patients unless the CD4+ count is ≥ 300/μL, viral load is undetectable, and the patient is currently receiving highly active antiretroviral therapy.

Exclusion Criteria: (Group A) A1. Patients previously exposed to afatinib. A2. History of interstitial lung disease (ILD), ILD-like adverse reactions (such as lung infiltration, pneumonitis, acute respiratory distress syndrome, allergic alveolitis), or radiation pneumonia requiring steroid therapy.

Exclusion Criteria: (Group B) B1. More than 2 lines of a second-generation hormonal agent for metastatic disease.

B2. More than 2 lines of systemic chemotherapy for metastatic disease. B3. Patients with only nonmeasurable lesions other than bone metastasis (eg, pleural effusion, ascites, other visceral locations). B4. A history of seizure or any condition predisposing patient to seizure within 12 months before study treatment, including history of unexplained loss of consciousness or transient ischemic attack, for patients receiving enzalutamide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of response. | Every 8 weeks until study ends, approximately 2 years
  Objective Response Rate (ORR) by local assessment per RECIST v1.1
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of Prostate-Specific antigen level ≥ 50% (PSA50) response. | Every 4 weeks until study ends, approximately 2 years
  PSA50 response rate

SECONDARY OUTCOMES:
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by local investigator | Every 8 weeks until study ends, approximately 2 years
  Objective Response Rate (ORR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by local investigator | Every 8 weeks until study ends, approximately 2 years
  Duration of Response (DOR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by local investigator | Every 8 weeks until study ends, approximately 2 years
  Time to Response (TTR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by independent central review | Every 8 weeks until study ends, approximately 2 years
  Objective Response Rate (ORR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by independent central review | Every 8 weeks until study ends, approximately 2 years
  Duration of Response (DOR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by independent central review | Every 8 weeks until study ends, approximately 2 years
  Time to Response (TTR) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by independent central review | Every 8 weeks until study ends, approximately 2 years
  Progression-free Survival (PFS) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of antitumor activity as assessed by local investigator | Every 8 weeks until study ends, approximately 2 years
  Progression-free Survival (PFS) per RECIST v1.1
Group A: Evaluate efficacy of zenocutuzumab in combination with afatinib in terms of survival | Continuous through study completion, up to 2 years
  Overall Survival (OS)
Group A: Evaluate safety and tolerability of zenocutuzumab in combination with afatinib | continuous through study completion, an average of 9 months
  Frequency and nature of adverse events (AEs) that are related to treatment as assessed by Common Terminology Criteria for AEs (CTCAE) version 5.0
Group A: Maximum plasma concentration [Cmax] of zenocutuzumab when given in combination with afatinib | 12 months
  Cmax
Group A: Characterize immunogenicity of zenocutuzumab. | 12 months
  Incidence of antidrug antibodies against zenocutuzumab
Group A: Area under the concentration versus time curve from time zero to time t [AUC0-t] of zenocutuzumab when given in combination with afatinib | 12 months
  AUC0-t
Group A: Area under the concentration versus time curve [AUC0-∞] of zenocutuzumab when given in combination with afatinib | 12 months
  AUC0-∞
Group A: Area under the concentration versus time curve [AUC0-∞] of afatinib when given in combination with zenocutuzumab | 12 months
  AUC0-∞
Group A: Area under the concentration versus time curve from time zero to time t [AUC0-t] afatinib when given in combination with zenocutuzumab | 12 months
  AUC0-t
Group A: Maximum plasma concentration [Cmax] afatinib when given in combination with zenocutuzumab | 12 months
  Cmax
Group A: Characterize immunogenicity of zenocutuzumab. | 12 months
  Serum titers of antidrug antibodies against zenocutuzumab
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of antitumor activity as assessed by local investigator. | Every 8 weeks until study ends, approximately 2 years
  Objective Response Rate (ORR) per RECIST v1.1
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of Prostate-specific antigen level ≥ 30% (PSA30) response. | Every 4 weeks until study ends, approximately 2 years
  PSA30 response rate
Group B: Evaluate efficacy zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of survival parameters | Continuous through study completion, up to 2 years
  Radiographic Progression Free Survival (rPFS) by local investigator per Prostate Cancer Clinical Trials Working Group 3 Modified Response Evaluation Criteria in Solid Tumors (PCWG3-modified RECIST) v1.1 and Overall Survival (OS)
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of antitumor activity as assessed by local investigator. | Every 8 weeks until study ends, approximately 2 years
  Duration of Response (DOR) per PCWG3-modified RECIST v1.1
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of antitumor activity as assessed by local investigator. | Every 8 weeks until study ends, approximately 2 years
  Time to Response (TTR) per PCWG3-modified RECIST v1.1
Group B: Evaluate efficacy of zenocutuzumab in combination with enzalutamide or abiraterone acetate in terms of Prostate-specific antigen level ≥ 30% (PSA30) response. | Every 8 weeks until study ends, approximately 2 years
  time to Prostate-specific antigen (PSA) progression per PCWG3-modified RECIST v1.1
Group B: Evaluate safety and tolerability of zenocutuzumab in combination with enzalutamide or abiraterone acetate. | continuous through study completion, an average of 6 months
  Frequency and nature of adverse events (AEs) that are related to treatment as assessed by Common Terminology Criteria for AEs (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - Florida Cancer Specialists, Lake Mary, Florida
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - University Hospitals - Seidman Cancer Center, Cleveland, Ohio
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No